CLINICAL TRIAL: NCT00883818
Title: Detection and Treatment Benefit of Microorganism (Chlamydia Trachomatis, Mycoplasma Hominis, Ureaplasma Urealyticum) in Overactive Bladder Patients
Brief Title: Microorganism in Overactive Bladder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-12-027
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-06

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Mycoplasma
MeSH Terms: conditions — Urinary Bladder, Overactive; Mycoplasma Infections | interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotics therapy (Experimental)
  Interventions: Drug: azithromycin, doxycycline

INTERVENTIONS:
Drug: azithromycin, doxycycline — azithromycin 1g once for women with positive cultures at baseline
  doxycycline 100 mg twice daily for 7 days for women with persistent infection after treatment of azithromycin 1g
  Other Names: azithromycin; doxycycline

SUMMARY:
The objective of this prospective study is to determine the incidence of mycoplasma in women with overactive bladder (OAB) symptoms and whether antibiotic therapy targeting these organisms is effective.

DETAILED DESCRIPTION:
Overactive bladder (OAB) syndrome is described as 'urgency, with or without urge incontinence, usually with frequency and nocturia' by the 2002 ICS Terminology Committee. A variety of medical conditions share the symptoms of OAB, and it is important to exclude these in the process of diagnosis. Urinary tract infection (UTI) is the most frequent alternative diagnosis. Even in patients considered to have interstitial cystitis, OAB is a high probability of diagnosis due to its insidious onset of irritative symptoms.For these reasons, ICS Terminology Committee stated that the term OAB can be used only if there is no proven infection or other obvious pathology.

Isolating causative organisms through urine culture plays a crucial role, but is likely to reveal a positive result in less than half of patients presenting with irritative symptoms. Even though ordinary bacteria are not cultured from these patients, there is some evidence to suggest that atypical organisms, such as genital mycoplasma, may be associated with OAB symptoms. For example, 48% of patients with chronic voiding symptoms showed positive cultures for Ureaplasma urealyticum and Mycoplasma hominis. In 91% of the patients with positive culture, symptom severity and frequency were improved after treatment. Another evidence for mycoplasmal involvement in OAB symptoms derives from the improvements in symptoms in more than two-thirds of patients complaining of persistent frequency and urgency after the use of doxycyline which is effective against U. urealyticum, M. hominis and Chlamydia trachomatis.

Mycoplasmas are the simplest micro-organisms regarded as true bacteria. They are highly pleomorphic parasites of humans and the absence of a cell wall has been used to distinguish mycoplasma and to place them taxonomically in the class Mollicutes.Mycoplasmas are not generally viewed as being highly virulent, although they usually manifest a predilection for particular host tissues, such as the urogenital or respiratory tracts. It is now being recognized that these organisms play a more important role in human infections than was previously thought. Its slow-growing, non-culturable nature enables them to establish chronic infections, resist the effects of antibiotics and protect the organisms against immune system reactivity.Accordingly, for patients presenting with irritative bladder symptoms, and especially whose first culture is negative, a further culture may be indicated to test specifically for Mycoplasma or Chlamydia infection.

ELIGIBILITY:
Inclusion Criteria:

1. Women age of 20 ≤ and ≤ 80 years
2. Symptoms of urinary frequency (≥8 micturitions per 24 hours) and urinary urgency (defined as a level of 3 to 5 in a 5 point urgency scale) at least one episode a day as verified by baseline micturition diary
3. Symptoms of overactive bladder, including, urgency, frequency, and/or urinary urge incontinence for more than 3 months
4. No proven ordinary bacteria on routine urine culture or gram stain
5. Positive for one of Mycoplasma homonis, Ureaplasma Urealyticum and Chlamydia trachomatis on urethral or cervical swab

Exclusion Criteria:

1. Neurogenic bladder
2. Indwelling catheter
3. PVR ≥ 150ml
4. Interstitial cystitis
5. History of radiation therapy on pelvic area or chemotherapy
6. unable to record voiding diary
7. Pregnancy
8. Other reasons according to investigator's opinion

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of positive cultures for M. hominis, U. urealyticum and C. trachomatis in women with OAB symptoms. | Baseline

SECONDARY OUTCOMES:
Reduction rate in urinary frequency after treatment in women with positive culture at baseline. | 2 weeks after treatment
Changes in mean urgency episodes, PPBC scores, BFLUTS questionnaire and PPTB after treatment in women with positive culture at baseline. | 2 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Inha University College of Medicine, Inchon
  - Kangnam St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Asan Medical Center, Ulsan College of Medicine, Seoul